CLINICAL TRIAL: NCT01936805
Title: ROsuvastatin LOading and Clinical Outcomes Trial
Acronym: ROLOCO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yuksek Ihtisas Hospital (Other)
Responsible Party: Principal Investigator, Serkan Cay, Associate Professor, Yuksek Ihtisas Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2173862
Record Dates: First submitted 2013-08-09; First posted 2013-09-06 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-09

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rosuvastatin (Active Comparator): A 40 mg loading dose of rosuvastatin was administrated 24 h before the PCI.
  Interventions: Drug: Rosuvastatin
- Control (Placebo Comparator): A loading dose of placebo was administrated 24 h before the PCI.

INTERVENTIONS:
Drug: Rosuvastatin — A 40 mg loading dose of rosuvastatin was administrated 24 h before the PCI.
  Arms: Rosuvastatin

SUMMARY:
The aim of the present study was to evaluate the effect of pre-procedural single high loading dose (40 mg) of rosuvastatin on the primary end-points of all cause mortality and composite of death or myocardial infarction from cardiovascular (CV) causes, target vessel revascularization (TVR), or stroke.

ELIGIBILITY:
Inclusion Criteria:

* statin-naive patients
* stable ischemic heart disease
* de novo lesions appropriate for PCI

Exclusion Criteria:

* current statin use
* statin allergic patients
* acute coronary syndromes
* lesions not appropriate for PCI
* refusal for participation
* statin quitting during follow- up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2008-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
all cause death and composite of death or myocardial infarction from CV causes, TVR, or stroke | 4 year

SECONDARY OUTCOMES:
all cause death | 4 year
composite of death or myocardial infarction from CV causes, TVR, or stroke | 4 year

CONTACTS AND LOCATIONS:
Locations (1):
- Yuksek Ihtisas Hospital, Ankara, Altindag, Turkey (Türkiye)